CLINICAL TRIAL: NCT06915129
Title: Galactooligosaccharides (GOS) Promote the Proliferation of Bifidobacteria and May be a Viable Management Strategy for Lactose Intolerance Symptoms
Brief Title: The Effect of Galactooligosaccharides (GOS) on the Gut Microbiota of Lactose Intolerance Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Responsible Party: Principal Investigator, Dave Dallas, Assistant Professor, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-2021-1044
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2022-07

CONDITIONS: Modulation of the Human Gut Microbiota by Prebiotic Galactooligosaccharides (GOS)

STUDY DESIGN:
Intervention Model Description: The experimental design was a completely randomized placebo-controlled clinical trial study, which consisted of a one-week screening period followed by a 3-week supplementation period and a 3 week-washout period
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Galactooligosaccharides group(GOS)) (Experimental): During the supplementation period, participants were instructed to consume twice daily (morning and evening) prebagged 5.2 g of galactooligosaccharide (GOS) which the participants were instructed to dissolve in 250 ml of water and consume either before or after meals.
  Interventions: Dietary Supplement: Prebiotic galactooligosaccharides (GOS)
- Control group (lactose group) (Placebo Comparator): During the supplementation period, participants were instructed to consume twice daily (morning and evening) prebagged 1 g of lactose which the participant was instructed to dissolve in 250 ml of water and consume either before or after meals.
  Interventions: Dietary Supplement: Prebiotic galactooligosaccharides (GOS)

INTERVENTIONS:
Dietary Supplement: Prebiotic galactooligosaccharides (GOS) — Galactooligosaccharides (GOSs) are a group of nondigestible oligosaccharides consisting of galactose units linked via glycosidic bonds to galactose, terminal glucose, or sucrose. The linkages are not digested by human and animal pancreatic or intestinal enzymes. Some recent papers reported that daily supplementation with prebiotic GOS to lactose-intolerant individuals altered the gut microbiome and decreased lactose intolerance (LI) symptoms.

SUMMARY:
The purpose of this study was to identify specific microbes that change with supplementation with galactooligosaccharides-prebiotics that are associated with alleviation of lactose intolerance symptoms in lactose-intolerant human subjects.

DETAILED DESCRIPTION:
The experimental design of this study was a completely randomized placebo-controlled clinical trial study, which consisted of a one-week screening period followed by a 3-week supplementation period and a 3 week-washout period. Institutional Review Board (IRB) approval was obtained through Oregon State University's Regional Institutional Review Board (IRB Number IRB-2021-1044) and written informed consent was obtained from all participants.

During the supplementation period, participants were instructed to consume twice daily (morning and evening) either prebagged 5.2 g of GOS (treatment group) or 1 g of lactose (placebo), which the participants were instructed to dissolve in 250ml of water and consume either before or after meals. The GOS (donated by FrieslandCampina, Amersfoort, the Netherlands, and sold under the trade name, BiotisTM GOS-O Powder) contained 73.7% GOS, 20.9% lactose, and 5.3% monosaccharides (galactose and glucose) and 1.0% ash. To account for the nutritional impact of lactose in the GOS supplement on host and microbiota, 1 g lactose, donated by Glanbia Nutritionals (Twin Falls, ID, USA), was given as a control in this study.

12 adults (2 males, 10 females), ages 19-55 years (mean: 29 years; SD: 11 years) started the clinical trial. During the study, participants continued with their regular diets that they recorded weekly in a food frequency questionnaire. The only dietary restrictions were: no consumption of dairy pills such as Lactaid, no pre/probiotic supplements, and antibiotics.

Fecal samples were collected weekly for the duration of the study. Participants used the Easy Sampler ® Stool Collection kit (ALPCO®, New Hampshire, USA) to collect samples and they dropped them off in the lab immediately after collection.

DNA was extracted from 200 mg of fecal samples via a QIAamp Powerfeccal Pro(Qiagen, Hilden, Germany).

The concentration of extracted DNA was measured via a Qubit 4 Fluorometer (Thermo Fisher Scientific, Waltham, MA) followed by a library construction targeting the V4 region of the 16S rRNA gene for microbiome sequencing.

Microbiome compositional analysis and statistical analysis were performed to identify shifts in specific microbes over time with prebiotic GOS supplementation and lactose supplementation.

Selected lactose-fermenting-related biomarker microorganisms were kept track of for any significant increases or decreases in relative abundance as well as any other microbes that have not been previously reported.

For the duration of the study, participants recorded gastrointestinal symptoms every other day in an unvalidated, online questionnaire which was specifically designed for this study to capture the incidence and severity of LI symptoms (abdominal pain, bloating, burping, constipation, diarrhea, discomfort during defecation, flatulence, heart burn, incomplete defecation, nausea, urgency to defecate).

To evaluate the impact of diet on microbial diversity and gastrointestinal symptoms, we correlated weekly food group intake with weekly measure of microbial diversity and gastrointestinal symptoms overall, within GOS, and within Control using Spearman correlation in SAS.

ELIGIBILITY:
Inclusion Criteria:

- People with lactose intolerance (formal and informal diagnosis) Fluent in English People who have a primary care provider Have to be 18 years and older

Exclusion Criteria:

- Any known gastrointestinal disease or disorder, or major gastrointestinal surgery Habitual use of laxatives or antacids Diabetes Pregnancy Use of antibiotics within one month prior to the study Use of pre or probiotics within one month prior to the study Any subject who, in the opinion of a physician, has a medical or psychological condition that would preclude them from completing the study Dairy protein allergy (not lactose intolerance) Use of lactose intolerance pills such as "Lactaid" should be avoided during the course of this study

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Increase in the relative abundance of the genus Bifidobacterium and other lactose-metabolizing genera | 6 weeks
  DNA was extracted from 200 mg of fecal samples Hilden, Germany). The concentration of extracted DNA was measured by Fluorometer, followed by a library construction targeting the V4 region of the 16S rRNA gene for microbiome sequencing.
  Microbiome compositional analysis and statistical analysis was performed to identify shifts in specific microbes over time with prebiotic GOS supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Milam Hall, Room 001, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided